CLINICAL TRIAL: NCT01814644
Title: Tailored Rapid Interactive Mobile Messaging (TRIMM) for Weight Control Among the Underserved
Brief Title: Interactive Mobile Messaging for Weight Control Among the Underserved
Acronym: TRIMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0003436
Record Dates: First submitted 2012-07-31; First posted 2013-03-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Individual assessment Lifestyle counseling
  Interventions: Behavioral: Standard Care
- TRIMM Intervention (Experimental): Individual assessment Lifestyle counseling Text messages
  Interventions: Behavioral: TRIMM Intervention

INTERVENTIONS:
Behavioral: TRIMM Intervention — Individuals in the TRIMM arm receive daily, individualized text-messages promoting positive lifestyle changes to support weight loss/management.
  Arms: TRIMM Intervention
Behavioral: Standard Care — Individual assessment, lifestyle counseling
  Arms: Standard Care

SUMMARY:
This project will test the efficacy of the "TRIMM" (Tailored Rapid Interactive Mobile Messaging) program, a user-friendly, semi-individualized text-messaging intervention to facilitate lifestyle change and weight loss among obese African-American adults with or at risk for diabetes, in a pilot, controlled clinical trial.

The text-messaging intervention will be in addition to, and compared with traditional diet, behavior, and physical activity education. Tips will be designed to increase knowledge, skills, and motivation.

DETAILED DESCRIPTION:
Type-2 diabetes, and its most important risk factor, obesity, have become major strains on our nation's health care system. By 2050, one in three U.S. adults could have diabetes (Stobbe, 2010), and obesity currently contributes nearly 17% of U.S. medical costs (Cawley, 2010). Our nation's underserved urban minority populations disproportionately suffer from type-2 diabetes and obesity. African-Americans, for example, comprise 12% of the US population but 23% of the extremely obese (Livingston, 2004). To reduce diabetes, obesity must be addressed. Unfortunately, traditional obesity interventions are intrusive and costly.

This project will test the efficacy of the "TRIMM" (Tailored Rapid Interactive Mobile Messaging) program, a user-friendly, semi-individualized text-messaging intervention to facilitate lifestyle change and weight loss among obese African-American adults with or at risk for diabetes, in a pilot, controlled clinical trial.

The text-messaging intervention will be in addition to, and compared with traditional diet, behavior, and physical activity education. Tips will be designed to increase knowledge, skills, and motivation. Participants will have the option to receive spiritually-based messages, if desired.

166 overweight or obese men and women will be recruited from 10 Baltimore inner-city churches, and will be assigned to one of two, six-month lifestyle-change programs. Participants must be overweight, aged 21-65, and own a cell phone with text-messaging capability. To be eligible for the study, participants will need to first pass a health screening and meet other study criteria.

The McKesson Foundation is funding this study, which has a total of 5 visits, ranging from ½ hr. to 3 hrs. The active intervention will last 6 months, with a follow-up visit at month 12. The TRIMM Program will feature periodic, individualized text messages and feedback via the participant's mobile phone as well as periodic follow-up appointments. The traditional program will consist of traditional diet, behavior, and physical activity education.

Qualified participants will receive individualized weight-loss plans and monetary compensation for their time, effort, & parking.

The long-term goal is to demonstrate, using a real-life setting, the potential superiority in efficacy of a specific mHealth application (text-messaging) for an underserved population at high risk of type-2 diabetes, compared to traditional, often more costly, and currently underutilized lifestyle-change interventions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be African-American,
* aged 21-65,
* have a phone with unlimited text/SMS capability,
* a BMI > 27, and
* be free from uncontrolled hypertension or other health or mental health condition that would make it inappropriate or unsafe for them to participate.

Exclusion Criteria:

* Following initial assessments, participants will be excluded if they are currently abusing alcohol/other substances, or
* have an Inventory of Depressive Symptomatology (IDS-SR) score > 38 ('severe to very severe' depression).

Potential participants with uncontrolled hypertension (> 160 systolic or >95 diastolic), HbA1c > 8, or symptomatic CAD will be referred for medical clearance.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Biometrics | Change from month 0 (baseline) to month 3, 6, and 12
  Physical measures: weight, blood pressure, resting heart rate, height, and waist circumference
Impact of Weight on Quality of Life | Change from month 0 (baseline) to month 6
  The Lite Version (IWQOL-Lite)is a widely used, well-validated, and reliable 31-item survey of obesity related quality of life (Kolotkin, 2002).
Diet quality | Change from month 0 (baseline) to month 6
  The 2005 Healthy Eating Index (HEI-2005) is a standardized tool that measures diet quality compared to MyPyramid.gov and the 2005 U.S. Dietary Guidelines. The 24-hour dietary recall is used to calculate the 12 components of the HEI-2005. HEI scores range from 0 to 100 (best) (USDA, 2000).
Nutrition knowledge and beliefs. | Change from month 0 (baseline) to month 6
  The 2008 Health and Diet Survey (HDS) will be used to assess participant's knowledge and attitudes, important components of the Health Belief Model. Questions cover nutrition knowledge and attitudes, grocery shopping, food label use, etc.
Exercise Benefits/Barriers | Change from month 0 (baseline) to month 6
  The Exercise Benefits/Barriers Scale (EBBS). This scale was developed to understand individuals' perceptions of the benefits of and barriers to participating in exercise.
Self-Efficacy for Exercise | Change from month 0 (baseline) to month 6
  The Self-Efficacy for Exercise Scale (SEE) is a 13-item measure that focuses on self-efficacy and expectations related to the ability to continue to exercise in the face of barriers.
Self-Efficacy for Weight Loss | Change from month 0 (baseline) to month 6
  Weight Efficacy Lifestyle Questionnaire (WEL). This will be used to assess self-efficacy for weight loss. The 20-item WEL consists of five situational factors: Negative Emotions, Availability, Social Pressure, Physical Discomfort, and Positive Activities.
Motivation/Readiness to Change | Change from month 0 (baseline) to month 6
  University of Rhode Island Change Assessment Scale. (URICA; McConnaughy, Prochaska, & Velicer, 1983). This will be used to assess motivation and readiness to change; based on the Transtheoretical Model of health behavior change. Accurately assessing motivation or commitment to change is a crucial step in matching patients to appropriate interventions.
Depression | Change from month 0 (baseline) to month 6
  The Inventory of Depressive Symptomatology: Self-Report. The DS-SR will be used to assess symptoms of depression (Rush, 1986, 1996). Its psychometric properties have been established in various populations (Rush 1996, 2000).
Barriers to Change | Change from month 0 (baseline) to month 6
  These will be examined using a measure specifically developed for use in this study. Barriers assessed in the survey were identified via a focus group with the target population, existing literature on lifestyle change programs, and the investigators prior experience conducting health behavior change interventions.

SECONDARY OUTCOMES:
Process survey | month 6
  Participants will be given a survey assessing intervention's ease of use, satisfaction and desire to continue use at 6 months to obtain process evaluation measures.

REFERENCES:
- [Derived] Lin M, Mahmooth Z, Dedhia N, Frutchey R, Mercado CE, Epstein DH, Preston KL, Gibbons MC, Bowie JV, Labrique AB, Cheskin LJ. Tailored, interactive text messages for enhancing weight loss among African American adults: the TRIMM randomized controlled trial. Am J Med. 2015 Aug;128(8):896-904. doi: 10.1016/j.amjmed.2015.03.013. Epub 2015 Mar 31. PMID 25840035